CLINICAL TRIAL: NCT07023744
Title: A Triple-Blind, Placebo-Controlled, Randomized Clinical Trial of CANnabinoids for Drug Resistant Epilepsy in Adults and Children
Brief Title: CANnabinoids for Drug Resistant Epilepsy (DRE) in Adults and Children
Acronym: CAN-DRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Research Manitoba (Other)
Responsible Party: Principal Investigator, Lauren Kelly, PhD, MSc, BMedSci, CCRP, Associate Professor, Dept. of Pediatrics & Child Health, University of Manitoba Scientific Director, the Canadian Collaborative for Childhood Cannabinoid Therapeutics (https://www.medcannkids.ca/), University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN-DRE
Record Dates: First submitted 2025-05-22; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Drug Resistant Epilepsy
Keywords: adult and children; cannabis; DRE; CBD-isolate; CBD-enriched Cannabis Herbal Extract (CHE); cannabidiol
MeSH Terms: conditions — Drug Resistant Epilepsy; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: an early phase, triple-blind, placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Placebo Arm (MPL-012) (Placebo Comparator): Placebo arm -> MPL-012 oil, each mL contains 0mg CBD and 0mg THC.
  Interventions: Drug: Placebo
- Arm 2 - CBD Isolate (MPL-015) (Experimental): CBD-Isolate arm -> MPL-015 oil, each ml contains 100mg CBD and 0mg THC.
  Interventions: Drug: CBD Isolate
- Arm 3 - CBD-CHE (MPL-016) (Experimental): CBD-CHE arm -> MPL-016 oil, a CBD-enriched cannabis herbal extract, each ml contains 100mg CBD and 3mg THC.
  Interventions: Drug: CBD CHE

INTERVENTIONS:
Drug: Placebo — Placebo arm: participants will receive Placebo MPL-012 oil only through the trial participation. MPL-012 is produced by MediPharm Labs, each mL contains 0mg CBD and 0mg THC.
  Arms: Arm 1 - Placebo Arm (MPL-012)
Drug: CBD Isolate — CBD Isolate: MPL-015 is a CBD isolate, produced by MediPharm Labs, each mL contains 100mg CBD and 0mg THC.
  Arms: Arm 2 - CBD Isolate (MPL-015)
Drug: CBD CHE — CBD-CHE arm: MPL -016 is a CBD-enriched cannabis herbal extract, produced by MediPharm Labs, each mL contains 100mg of CBD and 3mg of THC.
  Arms: Arm 3 - CBD-CHE (MPL-016)

SUMMARY:
Epilepsy is a neurological disorder affecting more than 50 million people globally, including more than 260,000 Canadians. Cannabidiol (CBD) reduces seizure frequency and improves quality of life for adults and children with Drug Resistant Epilepsy (DRE). Several uncontrolled, small, open label studies reported that CBD-enriched Cannabis Herbal Extract (CHE) resulted in a reduction of seizure frequency, but we lack critical information on efficacy, comparative effectiveness and dosing of CBD and ∆9-tetrahydrocannabinol (THC) in children and adults with DRE. CAN-DRE is an early phase, triple-blind, placebo-controlled, randomized clinical trial to answer the questions of if cannabinoids work to reduce seizures in children and adults (24 months to 55 years) with DRE and if CBD works better in an isolate or in a CBD-enriched Cannabis Herbal Extract. The primary outcome of CAN-DRE is reported monthly seizure count from baseline to maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 24 months to 55 years old at the time of enrollment
2. Diagnosed with DRE: not achieved seizure freedom, with adequate trials of 2 antiseizure medications 29
3. Medical history of 4 + clinically recognizable seizures (any type with clusters counted as a single event) per month
4. Have a negative pregnancy test at screening for patients who have experienced menarche
5. Agree to abstain from driving and recreational cannabis use throughout the study

Exclusion Criteria:

1. Diagnosis of psychogenic non-epileptic seizure
2. Recent (<30 days) change in anticonvulsant therapies including anticonvulsant medications, or settings on vagal nerve stimulator
3. Ketogenic diet started within 6 months (participants stable on the ketogenic diet for more than 6 months are eligible to participate)
4. Vagal nerve stimulator implanted and activated within 12 months
5. Concomitant regular use of narcotics (except in emergencies and physician supervised)
6. Initiation or dosage change of oral or injected steroids within 3 months
7. Allergy or intolerance to compounds in trial preparations
8. DRE secondary to progressive neurological disease
9. Clinically significant cardiac, renal or hepatic disease (as assessed by site investigator); elevated liver enzymes (GGT and/or AST and/or ALT) or lipase >3 times upper limit, adjusted for age
10. History of psychotic disorders
11. Uncontrolled (in the perspective of the qualified investigator) medical conditions including substance use disorders
12. History or concurrent cannabis use disorder
13. Unwilling or unable to use highly effective methods of contraception throughout the study period and three months post-trial, where applicable

Ages: 24 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy in reducing seizure frequency | 116 days
  reported monthly seizure count from baseline to maintenance
Cannabinoid-related AEs and DLTs | 116 + 60 days
  The frequency and type of adverse events and dose limiting toxicities (DLTs) reported by caregivers and participants throughout the trial participation

SECONDARY OUTCOMES:
participant/family acceptability of this trial design | 116 days
  to be measured via post-study questionnaire, open-ended questions asked, no specific scale is used.
Quality of Life reported by adult participant/family | 116 days
  Quality of Life in Epilepsy Inventory (QOLIE-31) tool for adult participants. Changes from baseline to maintenance phase will be compared to measure the outcome.
health resource utilization and changes | 176 days
  A trial-specific Health Resource Utilization Questionnaire (HRUQ) is used to collect epilepsy participants' healthcare resource usage and out-of-pocket healthcare expenses during trial participation. The data will be analyzed descriptively to measure direct and indirect healthcare resource utilization related to the intervention from baseline phase to 60-day follow up post study protocolized treatment.
changes in work and activity impairment affected by seizure | 116 days
  WPAI (Work Productivity and Activity Impairment Questionnaire) asks about the effect of participant's seizure on their/their caregivers' ability to work and perform regular activities. Changes reported from baseline to maintenance phase will be compared.
Quality of Life reported by pediatric participants and family | 116 days
  Quality of Life in Childhood Epilepsy (QOLCE-55) tool for pediatric participants (4 - 17 yrs). Changes from baseline to maintenance phase will be compared to measure the outcome.

IPD SHARING:
Plan to Share IPD: Undecided
No, summary level data may be available from the CAN-DRE steering committee following research ethics board approval.